CLINICAL TRIAL: NCT00559689
Title: Phase 4 Study of Once-Daily Inhaled Glucocorticosteroid Administration in Asthma Patients
Brief Title: Study of Inhaled Glucocorticosteroid Administration in Asthma Patients
Status: Completed | Type: Observational
Sponsor: Hamamatsu University (Other)
Other Study IDs: Hamamatsu-17-43; H-17-43
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: asthma patients; well-controlled
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: receive once-daily administration of inhaled glucocorticosteroids at bedtime
  Interventions: Drug: Budesonide,hydrofluoroalkane-beclomethasone
- 2: receive twice-daily administration of inhaled glucocorticosteroids
  Interventions: Drug: Budesonide,hydrofluoroalkane-beclomethasone dipropionate

INTERVENTIONS:
Drug: Budesonide,hydrofluoroalkane-beclomethasone dipropionate — receive twice-daily administration
  Groups: 2
Drug: Budesonide,hydrofluoroalkane-beclomethasone — once-daily administration at bedtime
  Groups: 1

SUMMARY:
Once-daily inhaled glucocorticosteroids treatment can sufficiently control airway inflammation in asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Receive ICS for one year or more, with no change in dose within the previous 8 weeks

Exclusion Criteria:

* Two or more courses of oral corticosteroid in the previous 12 months
* Admission to hospital due to asthma in the previous 6 months
* Admission to the intensive care unit due to asthma at any time in the past
* Current cigarette smoker.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Hospital
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2005-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
once-daily administration of inhaled glucocorticosteroids can control airway inflammation | two-year

CONTACTS AND LOCATIONS:
Overall Officials: Kingo Chida, MD,PhD, Study Chair
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan